CLINICAL TRIAL: NCT03296670
Title: Intracoronary Infusion of Alprostadil and Nitroglycerin With Targeted Perfusion Microcatheter in STEMI Patients With Coronary Slow Flow Phenomenon
Brief Title: Efficacy of Intracoronary Infusion of Different Medicine in STEMI Patients With CSFP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSG1501104
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2017-09

CONDITIONS: ST Segment Elevation Myocardial Infarction; Coronary Slow Flow Phenomenon
Keywords: STEMI; CSFP; Alprostadil; targeted perfusion microcatheter
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Alprostadil; Nitroglycerin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alprostadil (Experimental): alprostadil,2ug, delivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients with CSFP
  Interventions: Drug: Alprostadil
- nitroglycerin (Placebo Comparator): nitroglycerin,200ug, delivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients with CSFP
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Alprostadil — alprostadil,2ug, delivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients with CSFP
  Arms: alprostadil
Drug: Nitroglycerin — Nitroglycerin,200ug, delivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients with CSFP
  Arms: nitroglycerin

SUMMARY:
The study intends to evaluate the efficacy of different medicine delivering by targeted perfusion catheter in coronary administration on coronary blood flow in STEMI patients with CSFP.

DETAILED DESCRIPTION:
The goal of STEMI therapy is to successfully restore epicardial blood flow. PCI has been documented as being the most effective method for restoration of epicardial blood flow. However, stenting does not necessarily equate to epicardial blood flow; not every patient achieves TIMI 3 flow after successful PCI.

Currently, there are two main types of interventions to improve epicardial blood flow. One is the mechanical method, which included thrombus aspiration catheter and the distal protective devices. It has been confirmed that the mechanical method can effectively improve epicardial and myocardial perfusion in patient with part of large vessels and high burden thrombus. But for patients with small vessels and no obvious visual thrombus, the efficacy is not significant.

The other intervention is medicine which included GP IIb/IIIa receptor antagonist, adenosine, sodium nitroprusside, verapamil etc. Part of the drugs have some effect but the overall clinical efficacy is still not satisfied.

The study intends to use targeted perfusion catheter to deliver drug to the distal targeted blood vessels. TFG and cTFC are applied to evaluate the efficacy of treatment with Alprostadil or Nitroglycerin on coronary blood flow in STEMI patients with CSFP.

ELIGIBILITY:
Inclusion Criteria:

Patents with myocardial infarction who have symptom onset within 12h before randomization; ECG: ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads ; Corrected TIMI frame counted (cTFC) measured from the final angiographic imaging after PCI exceeding 40 frames; Signed informed consent form prior to trial participation.

Exclusion Criteria:

Coronary artery bypass surgery (CABG) history; Failed in stents implanting; Severe heart failure; Cardiogenic shock.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
TIMI Flow Grade (TFG) | One mins after PCI
  TIMI Flow Grade (TFG)assesses flow in the epicardial arteries
TIMI Flow Grade (TFG) | One mins after intracoronary medicine infusion post-PCI
  TIMI Flow Grade (TFG)assesses flow in the epicardial arteries
TIMI Frame Count (CTFC) | One mins after PCI
  CTFC is a continuous measurement assessing flow in the epicardial arteries.
TIMI Frame Count (CTFC) | One mins after intracoronary medicine infusion post-PCI
  CTFC is a continuous measurement assessing flow in the epicardial arteries.

SECONDARY OUTCOMES:
LVEF by echocardiography | Echocardiography was performed 3-7 days after PCI
  Echocardiographic index includes LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Ben He, MD,PhD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, China

REFERENCES:
- [Background] Ding S, Pu J, Qiao ZQ, Shan P, Song W, Du Y, Shen JY, Jin SX, Sun Y, Shen L, Lim YL, He B. TIMI myocardial perfusion frame count: a new method to assess myocardial perfusion and its predictive value for short-term prognosis. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):722-32. doi: 10.1002/ccd.22298. PMID 19960517
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Chinese Society of Cardiology of Chinese Medical Association; Editorial Board of Chinese Journal of Cardiology. [Guideline of non-ST segment elevation acute coronary syndrome]. Zhonghua Xin Xue Guan Bing Za Zhi. 2012 May;40(5):353-67. No abstract available. Chinese. PMID 22883082
- [Background] Kidambi A, Mather AN, Motwani M, Swoboda P, Uddin A, Greenwood JP, Plein S. The effect of microvascular obstruction and intramyocardial hemorrhage on contractile recovery in reperfused myocardial infarction: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jun 27;15(1):58. doi: 10.1186/1532-429X-15-58. PMID 23806080
- [Background] Roe MT, Ohman EM, Maas AC, Christenson RH, Mahaffey KW, Granger CB, Harrington RA, Califf RM, Krucoff MW. Shifting the open-artery hypothesis downstream: the quest for optimal reperfusion. J Am Coll Cardiol. 2001 Jan;37(1):9-18. doi: 10.1016/s0735-1097(00)01101-3. PMID 11153779
- [Background] Pu J, Shan P, Ding S, Qiao Z, Jiang L, Song W, Du Y, Shen J, Shen L, Jin S, He B. Gender differences in epicardial and tissue-level reperfusion in patients undergoing primary angioplasty for acute myocardial infarction. Atherosclerosis. 2011 Mar;215(1):203-8. doi: 10.1016/j.atherosclerosis.2010.11.019. Epub 2010 Nov 26. PMID 21176835
- [Background] Pu J, Ding S, Shan P, Qiao Z, Song W, Du Y, Shen J, Jin S, He B. Comparison of epicardial and myocardial perfusions after primary coronary angioplasty for ST-elevation myocardial infarction in patients under and over 75 years of age. Aging Clin Exp Res. 2010 Aug;22(4):295-302. doi: 10.1007/BF03337726. Epub 2009 Dec 1. PMID 20009495
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Shen LH, Wan F, Shen L, Ding S, Gong XR, Qiao ZQ, Du YP, Song W, Shen JY, Jin SX, Pu J, Yao TB, Jiang LS, Li WZ, Zhou GW, Liu SW, Han YL, He B. Pharmacoinvasive therapy for ST elevation myocardial infarction in China: a pilot study. J Thromb Thrombolysis. 2012 Jan;33(1):101-8. doi: 10.1007/s11239-011-0657-7. PMID 22094974
- [Derived] Sheng X, Ding S, Ge H, Sun Y, Kong L, He J, Pu J, He B. Intracoronary infusion of alprostadil and nitroglycerin with targeted perfusion microcatheter in STEMI patients with coronary slow flow phenomenon. Int J Cardiol. 2018 Aug 15;265:6-11. doi: 10.1016/j.ijcard.2018.04.119. Epub 2018 Apr 25. PMID 29728334